CLINICAL TRIAL: NCT02012075
Title: Efficacy and Safety Comparison of Extended-Release Carvedilol Sulfate and Sustained-release Metoprolol Succinate in Patients With Heart Failure
Brief Title: A Phase Ⅲ Study of Extended-Release Carvedilol Sulfate for the Treatment of Heart Failure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KWDLHF2012
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended-Release Carvedilol Sulfate (Experimental): 18-72mg/d,po
  Interventions: Drug: Extended-Release Carvedilol Sulfate
- Sustained-release Metoprolol Succinate (Active Comparator): 11.875-190mg/d,po
  Interventions: Drug: Sustained-release Metoprolol Succinate

INTERVENTIONS:
Drug: Extended-Release Carvedilol Sulfate
  Arms: Extended-Release Carvedilol Sulfate
Drug: Sustained-release Metoprolol Succinate
  Arms: Sustained-release Metoprolol Succinate

SUMMARY:
The aim of present study is to evaluate the efficacy and safety of Extended-Release Carvedilol Sulfate versus Sustained-release Metoprolol Succinate in Patients With Mild or Moderate Chronic Heart Failure.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females
* Aged from 18 to 75 years
* New York Heart Association(NYHA) classification Ⅱ-Ⅲ
* At screening, subject has an LVEF<0.45
* Have received optimal therapy with an Angiotensin converting enzyme inhibitors or angiotensin receptor blocker for 4 weeks before enrollment
* Subjects with symptoms of Stable heart failure do not need intravenous injection diuretics,cardiac inotropes or vasodilators
* Willing to provide written informed consent

Exclusion Criteria:

* Current treatment on any Class I or III antiarrhythmic, except amiodarone or beta-blockers
* Current treatment on calcium antagonists except for long-acting dihydropyridine agents
* Have a history of acute coronary syndrome,cerebral apoplexy or transient ischemic attack with 3 months
* Have a history of cardio-vascular surgery or other vessel operations with 3 months
* Have a history of sustained ventricular tachycardia or ventricular fibrillation with 3 months
* Have a plan to receive coronary revascularization or heart transplantation
* Uncontrolled ventricular arrhythmias (not controlled with antiarrhythmic therapy or an implantable defibrillator)
* Subjects with uncorrected primary obstructive or severe regurgitative valvular disease，nondilated (restrictive) or hypertrophic cardiomyopathy
* Sitting systolic blood pressure≤90mmHg (based on an average of 3 readings)
* Current decompensated heart failure
* Second or third degree heart block，or sick sinus syndrome，a pacemaker is not placed
* Contraindication to vasodilators
* Have a history of cardiac resynchronization therapy or
* Have received cardioverter defibrillator or pacemaker with 1 month
* Resting heart rate<50 beats per minute(based on the average of 3 readings)
* Elevated liver enzymes (alanine aminotransferase or aspartate aminotransferase levels greater than 3 times upper limit of normal)
* Serum creatinine levels greater than 2 times upper limit of normal
* Current clinical evidence of obstructive pulmonary disease (e.g., asthma or bronchitis) requiring inhaled or oral bronchodilator or steroid therapy
* History of drug sensitivity or allergic reaction to alpha or beta-blockers
* Contraindication or intolerance to beta-blockers
* Pregnant or lactating women and women planning to become pregnant
* Has any systemic disease, including cancer, with reduced life expectancy (<12 months)
* Use of an investigational drug within 30 days of enrollment
* Participation in an investigational device trial within 30 days of enrollment
* Known drug or alcohol abuse 1 year prior to enrollment
* Has a history of psychological illness/condition that interferes with ability to understand or complete requirements of the study
* In the opinion of the investigator the subject is known to be noncompliant with prescribed medication regimen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in left ventricular ejection fraction(LVEF) by ultrasound cardiogram | Baseline and Week 36

SECONDARY OUTCOMES:
Change From Baseline in Left Ventricular End Systolic Volume Index | Baseline and Week 36
Change From Baseline in Left Ventricular End Diastolic Volume Index | Baseline and Week 36
Incidence of Hospitalizations From Exacerbation of Heart Failure | Baseline and Week 36
Incidence of Hospitalizations From All Causes | Baseline and Week 36
Incidence of Deaths From All Causes | Baseline and Week 36
Change From Baseline in New York Heart Association（NYHA）classification | Baseline and Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Professor, Principal Investigator — Beijing Anzhen Hospital
Locations (12):
- China (12):
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Tongji Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Taizhou Hospital, Taizhou, Zhejiang
  - Beijing ANZHEN Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Xuan Wu Hospital affiliated to Capital Medical University, Beijing
  - Beijing Tongren hospital affiliated to Capital Medical University, Beijing